CLINICAL TRIAL: NCT00156260
Title: UMCC 2-48 Feasibility Study of Evaluating Breast Cancer Patients With Ductal Lavage
Brief Title: Feasibility Study of Evaluating Breast Cancer Patients With Ductal Lavage
Status: Terminated | Type: Observational
Sponsor: University of Michigan Rogel Cancer Center (Other)
Other Study IDs: UMCC 2-48
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2008-10-08 (Estimated); Status verified 2008-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Procedure: Ductal lavage

SUMMARY:
The primary purpose of this research is to analyze the cells present in the fluid obtained via ductal lavage from the nipple of a woman with a known diagnosis of breast cancer. A portion of the lavage fluid may be used in future breast cancer biomarkers. Remaining lavage fluid will be used to analyze its biochemical composition, for investigational purposes only.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age
2. biopsy-proven unilateral invasive breast cancer of any histology or ductal carcinoma in situ
3. patient desires or requires treatment with mastectomy
4. any patient who has undergone prior excisional biopsy of their primary breast tumor must have had margins positive for disease, or must have either mammographic or ultrasonographic evidence of probable residual disease in the breast.
5. patients receiving induction chemotherapy remain eligible for participation in the study regardless of tumor response; those with a clinical complete response remain eligible.
6. voluntarily signed informed consent. -

Exclusion Criteria:

1. male gender
2. lobular carcinoma in situ as the only cancerous histology
3. prior margin-negative excisional biopsy of primary breast tumor, with no evidence of residual disease
4. patient being treated with breast conservation therapy inability to understand the nature of the procedure pregnancy and/or active lactation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2003-01; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Newman, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Cancer Center, Ann Arbor, Michigan, United States